CLINICAL TRIAL: NCT05327764
Title: Work-To-Rest Ratios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Assistant Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006115
Record Dates: First submitted 2022-03-26; First posted 2022-04-14 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Randomized counterbalanced study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40:20 (Active Comparator): Walking for 40 minutes, resting for 20
  Interventions: Other: Work to rest cycles of 40:20 minutes
- 20:10 (Experimental): Walking for 40 minutes, resting for 20
  Interventions: Other: Work to rest cycles of 20:10 minutes

INTERVENTIONS:
Other: Work to rest cycles of 40:20 minutes — Walking in a hot environment for 2 hours with repeated 40 minutes of work and 20 minutes of rest
  Arms: 40:20
Other: Work to rest cycles of 20:10 minutes — Walking in a hot environment for 2 hours with repeated 20 minutes of work and 10 minutes of rest
  Arms: 20:10

SUMMARY:
The purpose of the study is to compare physiological responses to two hours of work adhering to two variations of a work-to-rest ratio in a hot environment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18-39 year old individuals
* Physically active

Exclusion Criteria:

* History of cardiovascular, metabolic, respiratory, neural, or renal disease
* Hypertensive or tachycardic during the screening visit (systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg, resting heart rate ≥ 100 bpm)
* Taking medication or supplements with a known side effect of affecting physiologic responses to exercise (e.g., acetaminophen, beta blockers, statins, aspirin)
* Any form of tobacco or nicotine use in the past six months
* Current musculoskeletal injury impacting physical activity
* A positive pregnancy test at any point in the study
* Study physician discretion based on any other medical condition or medication

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Change in core body temperature | Upon completion of 2 hours of the work protocol
  Core body temperature is measured using a rectal thermistor
Change in heart rate | Upon completion of 80 minutes of work
  Heart rate is measured using a telemetry strap

CONTACTS AND LOCATIONS:
Overall Officials: Riana Pryor, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share these data with other researchers.